CLINICAL TRIAL: NCT04810325
Title: Electrophysiologic Brain Sensing Using Implanted DBS Systems in Neurological and Psychiatric Disorders
Brief Title: Brain Sensing in Neurological and Psychiatric Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 296010
Record Dates: First submitted 2021-03-01; First posted 2021-03-22 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Movement Disorders; Dystonia; Parkinson Disease; Tremor
MeSH Terms: conditions — Movement Disorders; Dystonia; Parkinson Disease; Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
High-frequency deep brain stimulation (DBS) is an effective treatment strategy for a variety of movement disorders including Parkinson's disease, dystonia and tremor1-5, as well as for other neurological and psychiatric disorders e.g. obsessive compulsive disorder, depression, cluster headache, Tourette syndrome, epilepsy and eating disorders6-11. It is currently applied in a continuous fashion, using parameters set by the treating clinician. This approach is non-physiological, as it applies a constant, unchanging therapy to a dysfunctional neuronal system that would normally fluctuate markedly on a moment-by moment basis, depending on external stressors, cognitive load, physical activity and the timing of medication administration.

Fluctuations in physical symptoms reflect fluctuations in brain activity. Tracking and responding in real-time to these would allow personalised approaches to DBS through stimulating at appropriate intensities and only when necessary, thereby improving therapeutic efficacy, preserving battery life and potentially limiting side-effects12. Critical to the development of such adaptive/closed-loop DBS technologies is the identification of robust signals on which to base the delivery of variable high-frequency deep brain stimulation.

Local field potentials (LFPs), which are recordable through standard DBS electrodes, represent synchronous neuronal discharges within the basal ganglia. Different LFP signatures have been identified in different disorders, as well as in different clinical states within individual disorders. For example, low frequency LFPs in the Alpha/Theta ranges (4-12Hz) are frequently encountered in patients with Dystonia13,14, while both beta (12-30Hz) gamma (60-90Hz) band frequencies may be seen in Parkinson's disease, when the patient is OFF and dyskinetic, respectively15,16. Equally, suppression of these abnormal basal ganglia signals through medication administration or high-frequency DBS correlates with clinical improvement. As such, they represent attractive electrophysiologic biomarkers on which to base adaptive DBS approaches.

Until recently, neurophysiological assessments were purely a research tool, as they could only be recorded either intra-operatively or for a short period of time post-operatively using externalised DBS electrodes. However, advances in DBS technology now allow real-time LFP recordings to be simply and seamlessly obtained from fully implanted DBS systems e.g. Medtronic Percept PC.

In this study, we will evaluate a cohort of patients with movement disorders and other disorders of basal ganglia circuitry who have implanted DBS systems. Recordings of LFPs and/or non-invasive data such as EEG, limb muscle activation and movement (surface EMG and motion tracking) under various conditions (e.g. voluntary movement, ON/OFF medications, ON/OFF stimulation) will allow us to evaluate their utility as markers of underlying disease phenotype and severity and to assess their potential for use as electrophysiological biomarkers in adaptive DBS approaches. These evaluations in patients with DBS systems with and without LFP-sensing capabilities will take place during a single or multi-day evaluation (depending on patient preference and researcher availability). This study will advance not only the understanding of subcortical physiology in various disorders, but will also provide information about how neurophysiological and behavioural biomarkers can be used to inform personalised, precision closed-loop DBS approaches.

DETAILED DESCRIPTION:
Both hyperkinetic and hypokinetic movement disorders are associated with abnormal spatiotemporal activity within the basal ganglia circuitry13,16,17. This can be assessed through measuring local field potentials (LFPs), which represent the product of synchronous neuronal activity at a given site (unsynchronized, random activity being essentially cancelled out)13. Numerous other disorders such as obsessive compulsive disorder, major depression, Tourette's syndrome, epilepsy, eating disorders and cluster headaches are also amenable to successful modulation using DBS6-11. These disorders likely also have unique, disease-specific electrophysiological signatures, the exact nature of which remains to be thoroughly defined. Abnormal electrophysiological activity is useful not only in delineating the pathophysiologic underpinnings of these disorders, but is central to the future development of adaptive DBS systems which respond in real-time to ameliorate pathological brain acticity12. Adaptive DBS may provide further clinical benefit beyond currently employed continuous DBS approaches, with only a fraction of the energy requirements12.

Studies using microelectrode recordings at the time of DBS lead placement as well as recordings from externalised DBS electrodes have identified distinct neurophysiological signatures within different disorders. Examples include excess beta-frequency oscillations in Parkinsonism, alpha and theta frequency oscillations in dystonia and gamma oscillations in dyskinesia. These neurophysiologic biomarkers of disease can be affected by the application of high-frequency DBS. Future closed-loop DBS systems may rely on real-time suppression of such abnormal basal ganglia activity.

LFPs in Parkinson's disease

A significant body of work has confirmed that beta-frequency oscillations, recorded from both the subthalamic nucleus and the internal portion of the globus pallidus, correlate with severity of bradykinesia and rigidity in Parkinson's disease13,16-18. These beta-frequency oscillations are coherent across simultaneous recordings in different nuclei of the same patient, implying that these represent a network-level dysfunction in Parkinson's disease16,19. The amplitude/power of abnormal beta-frequency LFPs correlates with the severity of motor impairment in Parkinson's disease15,18. Moreover, beta-frequency LFPs can be suppressed both by levodopa administration, or by the application of high-frequency DBS20,21; in both scenarios the degree of suppression in beta-oscillations correlates with the degree of clinical motor improvement. Beta oscillations may therefore represent an electrophysiological parkinsonian symptom correlate which can act as a biomarker of the motor state. Hence, they may be useful signals on which to base stimulation using adaptive DBS technologies. However, some observations, such as the suppression of beta frequency oscillations during periods of tremor, have cast doubt on the robustness of this potential biomarker.

Other LFP frequency alterations have also been observed to correlate with clinical symptomatology in PD. For instance, synchronisation at frequencies in the gamma range (60-90Hz) have been correlated with dyskinesia, as have synchronisation at lower frequencies (4-8Hz)22,23. High-frequency oscillations in the 250Hz range have also been found to associate with parkinsonian clinical states and to shift to even higher frequencies (350Hz) following levodopa administration24. In contrast to beta-frequencies, changes in high-frequency LFPs do appear to correlate with tremor25.

Aside from pure frequency characteristics, the temporal distribution of beta-frequency oscillations has also been examined in different disease states. It is suggested that prolonged periods of beta synchronisation (beta bursts) may be responsible for the overall increase in beta power in patients with Parkinson's disease in the OFF state, and that a move to shorter durations of synchronisation may occur in the ON state26.

LFPs in dystonia

Patients with dystonia display a distinct pattern of LFP alterations in the pallidum13,14, particularly an excess of synchronized oscillatory activity in the low frequency 3-12 Hz band13. Not only is pallidal LFP power prominent in the 3-12Hz band in patients with dystonia13,27 but it correlates with28 and may be coherent with (especially contralateral) dystonic muscular activity29. Moreover, there is a direct association between pallidal low-frequency oscillations and dystonia severity30.

Increased LFP power in the low-frequency band is seen across a variety of dystonia phenotypes. In cervical dystonia, inter-hemispheric differences in LFPs have been demonstrated, though clear correlations with directional head movements have not been established31,32. In myoclonus-dystonia patients, increased pallidal LFP in the 3-15Hz range correlate with dystonic muscle activity33. Oscillatory activity may be different in secondary or combined dystonia, and may also differ according to genetic makeup 34-36.

LFPs in essential tremor

LFP recordings from patients undergoing thalamic DBS in ET have identified distinct thalamic LFP frequency characteristics, often coherent with surface EMG recordings in these groups, at frequencies which are either harmonics or subharmonics of the tremor frequency37.

LFPs in other conditions Electrophysiologic recordings from patients with Tourette's syndrome have shown an excess of low-frequency activity(2-13Hz) in both thalamic and pallidal targets38 and that spontaneous tics in Tourette's syndrome are preceded by coherent thalamo-cortical discharges39. Unique, disease specific LFP patterns have also been identified in a number of neuropsychiatric disorders. For example, prominent alpha activity in the basal ganglia has been suggested as an electrophysiologic correlate of major depressive disorders40

Continuous recording from fully implanted DBS systems has only recently become possible, for example using the Medtronic Percept PC battery system. The quality of signals recorded using this system as well as the correlation with clinical features, and coherence with cortical and motor activity however remain largely unexplored. Moreover, the number of patients on which previous LFP studies has been based is small. Hence, their utility in the future development of closed-loop DBS systems remains uncertain.

Our study will address a number of unanswered questions relating to the utility of LFP recordings in neurological disorders including:

1. Is it possible to replicate the previous findings concerning LFP signatures in various movement disorders using currently available DBS systems with LFP sensing capabilities e.g. Medtronic Percept PC?
2. Do LFP signatures persist many years after initiation of deep brain stimulation (most previous studies have evaluated patients only at the time of DBS implantation)?
3. How are LFP signatures related to modulations of wider brain networks as assessed by EEG?
4. Can non-invasive recording methods such as EEG provide alternative or complementary biomarkers for closed-loop DBS?
5. What is the influence of medications, body movements, sensory inputs and differential stimulation parameters on LFPs?
6. How robust are LFP signatures within and between individuals with similar disease states?
7. Do robust LFP signatures exist for non movement disorder basal ganglia network pathologies, and how do these correlate with symptoms severity?

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Neurological or psychiatric disorder treated with a DBS system.
* Able to give informed consent

Exclusion Criteria:

* • Inability to tolerate OFF stimulation conditions.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with neurological disorders treated with deep brain stimulation devices capable of neurophysiologic recording
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
local field potential power (amplitude) | 12 months
local field potential frequency (Hz) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Limousin, PhD, Principal Investigator — UCL

IPD SHARING:
Plan to Share IPD: Undecided